CLINICAL TRIAL: NCT02470988
Title: How is Psychological Change Experienced by Individuals Receiving Cognitive Behaviour Analysis System of Psychotherapy (CBASP) and How is This Affected by Disciplined Personal Involvement? A Multiple Baseline Single Case Design
Brief Title: Does Disciplined Personal Involvement Precede Change in CBASP?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15/WS/0027
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Chronic Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBASP (Active Comparator): Cognitive Behavioural Analysis System of Psychotherapy (CBASP) is a form of therapy specifically designed to treat individuals with chronic depression. CBASP combines a number of elements, with a focus on teaching the client to become aware of their interpersonal behaviour and its consequences.
  Interventions: Behavioral: Cognitive Behavioural Analysis System of Psychotherapy
- CBASP Without DPI (Experimental): In this arm CBASP will be delivered without Disciplined Personal Involvement (DPI) by the therapist.
  Interventions: Behavioral: CBASP Without DPI

INTERVENTIONS:
Behavioral: Cognitive Behavioural Analysis System of Psychotherapy
  Other Names: CBASP
  Arms: CBASP
Behavioral: CBASP Without DPI
  Arms: CBASP Without DPI

SUMMARY:
The purpose of the study is to investigate the process of symptom change in Cognitive Behavioural Analysis System of Psychotherapy (CBASP), and how the individual components of the therapy affect this change in individuals with chronic depression.

DETAILED DESCRIPTION:
A form of psychotherapy called Behaviour Analysis System of Psychotherapy (CBASP) has been developed specifically to treat individuals suffering from chronic, long-standing depression. There is a growing evidence base to suggest that CBASP is effective for these individuals, especially when combined with anti-depressant medication. This evidence comes from case series and randomised controlled trials that have compared CBASP with other forms of therapy such as Interpersonal Psychotherapy and Cognitive Behaviour Therapy, and with medication. The evidence from these studies consistently shows CBASP to be effective, and it compares favourably with other forms of therapy.

Given these findings, it is important to understand how change happens in CBASP and how it is affected by the components of the therapy. Understanding how individuals experience change within CBASP will have important implications for how the therapy is delivered in the future. For example if change is found to be non-linear it would be important to understand what components of the therapy are associated with improvement. There could also be organisational implications, for example relating to the optimal number of sessions to offer in order to achieve acceptable change while balancing therapist time.

The proposed study aims to investigate the process of psychological change in CBASP. This will be done by providing CBASP to a small number of individuals and gathering outcome data (rating of mood) at every therapy appointment. Session--by-session change will then be mapped for each participant. The study will include two arms: CBASP; and CBASP without Disciplined Personal Involvement (DPI). DPI involves specifically using the therapist--client relationship to help the client to discriminate between previous maladaptive relationships and other, positive ones. The reason for including this condition is to investigate whether DPI affects the process of psychological change in CBASP, as it is a unique feature of the therapy.

The study will use a single-case design, as the aim is to map change within each individual participant in the context of the therapy. This design was deemed appropriate as the study does not aim to make claims about the overall effectiveness of CBASP, but to provide an analysis of individual psychological change for participants receiving CBASP.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 64 years, inclusive
* Have been depressed for 2 years or longer
* Have had previous episodes of depression
* Previous treatment (medication, psychotherapy or both) unsuccessful or participant has relapsed
* Do not meet any of the exclusion criteria
* Able to provide informed consent to participate in the study

Exclusion Criteria:

* Received psychological therapy in previous 12 months
* Current significant substance misuse
* Presence of learning difficulties
* Presence of psychosis
* Unable to commit to the full duration of the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire - 9 (PHQ-9) | 6 months
  Administered at three weekly baseline assessments and then at every therapy session for all participants over a period of 6 months or up to 20 sessions.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - NHS Tayside, Dundee
  - NHS Lothian, Edinburgh